## NCT07211698

## A QUALITATIVE STUDY EXPLORING ETHNIC MINORITIES' EXPERIENCES OF HEALTHCARE INTERVENTIONS DELIVERED AT HOME OR IN COMMUNITY CENTRES

Ethnic Minorities' Experiences of Healthcare Intervention

18 JANUARY 2026





## INFORMED CONSENT FORM (for Individuals Delivering Falls Prevention Intervention in the Community)

Version 1.0, 18.01.2026

Short Study Title: Ethnic Minorities' Experiences of Healthcare Intervention

**REC Project ID:** FMHS 212-0725

Name of Chief Investigator: Dr Katie Robinson Name of PhD Researcher: Mrs Joy Watterson

| | | | Participant ID: | |
|---|---|---|---|---|
| | | | Please in | itial box |
| 1. | | | formation sheet version number 1.0 ad the opportunity to ask questions. | |
| 2. | | | nd that I am free to withdraw at any y medical care or legal rights being | |
| 3. | individuals from the Universal authorities where it is relevant individuals to have access | ersity of Nottingham,<br>ant to my taking part in<br>to these records and<br>ny participation in this | dy may be looked at by authorised the research group and regulatory this study. I give permission for these to collect, store, analyse and publish study. I understand that my personal | |
| 4. | I understand that the intervieus the interview may be used i | | nd that anonymous direct quotes from d PhD thesis. | |
| <ol><li>I understand that my contact information held and maintained by the research team may<br/>be used to help contact me or provide information about study findings.</li></ol> | | | | |
| <ol> <li>I understand that the information collected about me may be used to support<br/>other research in the future and may be shared anonymously with other researchers.</li> </ol> | | | | |
| 7. | I agree to take part in the al | bove study. | | |
| Name | of Participant | Date | Signature | |
| Name | of Person taking consent | Date | <br>Signature | |

**Governance Team Use Only - DO NOT DELETE** 



## Version Control and Revisions History Document title Consent Form (Qualitative Studies) Security Classification: Non-Confidential (Other UoN Staff) Document Review Due Date: 31-JAN-2027

Document Author: Kimberly Byrne

Document Owner Ali Alshukry

Responsible Team: Research Governance

Printed copies are uncontrolled

| Version | Date | Amendment | Made by |
|---|---|---|---|
| V1.1 | 11-JUL-2024 | Previous version | Kimberly Byrne |
| V1.2 | 15-OCT-2025 | Version control applied to existing document. Clause 2 updated in response to GDPR transparency wording update. Clause 6 updated | Kimberly Byrne |